CLINICAL TRIAL: NCT03000348
Title: A Randomized, Double-Blind, Parallel Group, Placebo-Controlled Study Investigating the Optimal Dose Regimen, Efficacy, and Safety of Adding Oral Cysteamine in Adult Patients Being Treated for an Exacerbation of CF-associated Lung Disease
Brief Title: A Study of the Dosing, Efficacy, and Safety of Oral Cysteamine in Adult Patients With Cystic Fibrosis Exacerbations
Acronym: CARE-CF1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NovaBiotics Ltd. (Industry)
Collaborators: Agility Clinical, Inc. (Industry); PSR Group B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NBTCS02
Record Dates: First submitted 2016-12-11; First posted 2016-12-22 (Estimated); Results first posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Cystic Fibrosis
Keywords: Exacerbation; CF; Lung disease; Lung infection; Gram negative; Bacterial Infection; pneumonia; bronchitis
MeSH Terms: conditions — Cystic Fibrosis; Lung Diseases; Bacterial Infections; Pneumonia; Bronchitis | interventions — Cysteamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- High Dose, Once per day (Active Comparator): Patient takes one oral dose of Cysteamine (high dose) per day, in the morning. The patient takes two oral placebo doses, one at mid-day and one in the evening.
  Interventions: Drug: Cysteamine; Drug: Placebo Oral Capsule
- High Dose, Twice per day (Active Comparator): Patient takes two oral doses of Cysteamine (high dose) per day, one in the morning and one in the evening. The patient takes one oral placebo dose, at mid-day.
  Interventions: Drug: Cysteamine; Drug: Placebo Oral Capsule
- High Dose, Three times per day (Active Comparator): Patient takes three oral doses of Cysteamine (high dose) per day, one in the morning, one at mid-day and one in the evening.
  Interventions: Drug: Cysteamine
- Placebo (Placebo Comparator): Patient takes three oral doses of placebo, one in the morning, one at mid-day and one in the evening.
  Interventions: Drug: Placebo Oral Capsule
- Low Dose, Three times per day (Active Comparator): Patient takes three oral doses of Cysteamine (low dose) per day, one in the morning, one at mid-day and one in the evening.
  Interventions: Drug: Cysteamine; Drug: Placebo Oral Capsule
- Mid-Range Dose, Three times per day (Active Comparator): Patient takes three oral doses of Cysteamine (mid-range dose) per day, one in the morning, one at mid-day and one in the evening.
  Interventions: Drug: Cysteamine; Drug: Placebo Oral Capsule

INTERVENTIONS:
Drug: Cysteamine — Oral Cysteamine Capsule
  Other Names: Lynovex; NM001; Lynovex Oral
  Arms: High Dose, Once per day; High Dose, Three times per day; High Dose, Twice per day; Low Dose, Three times per day; Mid-Range Dose, Three times per day
Drug: Placebo Oral Capsule — Placebo Oral Capsule
  Arms: High Dose, Once per day; High Dose, Twice per day; Low Dose, Three times per day; Mid-Range Dose, Three times per day; Placebo

SUMMARY:
This study investigates the use of cysteamine in the treatment of adults with Cystic Fibrosis who are experiencing an exacerbation of CF-associated lung disease. There are six different potential dosing regimens, including one that is placebo.

DETAILED DESCRIPTION:
This is a multicenter, double-blind, randomized, placebo-controlled, 6-arm study to investigate the optimal dose regimen, efficacy, and safety of cysteamine in the treatment of adult patients with CF who are experiencing an exacerbation of CF-associated lung disease. Patients will be screened for the study and eligible patients will be randomized to receive either cysteamine or placebo as add-on therapy to their standard of care treatment for CF-associated lung disease.

ELIGIBILITY:
Inclusion Criteria:

1. CF-associated lung disease with documented history of chronic infection with Gram-negative organism(s)
2. Established patient of the Principal Investigator's CF Multi Disciplinary Team (MDT)
3. Age ≥18 years
4. Weight >40 kg
5. FEV1 >30% of predicted within the 6 months prior to study exacerbation
6. At the baseline visit: experiencing a new exacerbation of CF-associated lung disease (based on Investigator assessment of ≥4 symptoms present on the Fuchs' criteria) requiring treatment that includes an aminoglycoside antibiotic
7. Females of childbearing potential will be included if they are either sexually inactive (sexually abstinent for 14 days prior to the first study drug dose continuing through 28 days after the last study drug dose, or using one of the following highly effective contraceptive (i.e. results in <1% failure rate when used consistently and correctly) methods in this trial:

   1. intrauterine device (IUD);
   2. surgical sterilization of the partner (vasectomy for 6 months minimum);
   3. combined (estrogen or progestogen containing) hormonal contraception associated with the inhibition of ovulation (either oral, intravaginal, or transdermal);
   4. progestogen only hormonal contraception associated with the inhibition of ovulation (either oral, injectable, or implantable);
   5. intrauterine hormone releasing system (IUS);
   6. bilateral tubal occlusion.
8. Females of childbearing potential agree to remain sexually inactive or to keep the same birth control method for at least 28 days following the last dose.
9. A female of non-childbearing potential must have undergone one of the following sterilization procedures at least 6 months prior to the first study drug dose:

   1. hysteroscopic sterilization;
   2. bilateral tubal ligation or bilateral salpingectomy;
   3. hysterectomy;
   4. bilateral oophorectomy; or be postmenopausal with amenorrhea for at least 1 year prior to the first study drug dose and follicle stimulating hormone (FSH) serum levels consistent with postmenopausal status.
10. A non-vasectomized male subject agrees to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days beyond the last dose of study medication and the female partner agrees to comply with inclusion 7 or 9. For a vasectomized male who has had his vasectomy 6 months or more prior to study start, it is required that they use a condom during sexual intercourse. A male who has been vasectomized less than 6 months prior to study start must follow the same restrictions as a non-vasectomized male.
11. If male, agrees not to donate sperm from the first study drug dose until 90 days after dosing.
12. Willing and able to comply with all protocol requirements and procedures, including induction of sputum, if necessary
13. Willing and able to provide signed and dated informed consent

Exclusion Criteria:

1. Hypersensitive to cysteamine or to any of the excipients
2. Hypersensitive to penicillamine
3. Transplant recipient
4. Participation in any other interventional clinical research study (participation in observational studies is not exclusionary) within 30 days of Baseline (Day 0), and any planned participation in an interventional clinical research study for the duration of this study
5. If female, pregnancy, planned pregnancy, or breast-feeding
6. Any other significant disease/disorder which, in the Investigator's opinion, either puts the patient at risk due to study participation, or may influence the results of the study or the patient's ability to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2016-12; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (8):
  - Banner University of Arizona Medical Center, Tucson, Arizona
  - San Francisco Critical Care Medical Group California Pacific Medical Center, San Francisco, California
  - University of Florida, Gainesville, Florida
  - Central Florida Pulmonary, Orlando, Florida
  - Albany Medical College, Albany, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - West Virginia University, Morgantown, West Virginia
  - The Medical College of Wisconsin/Froedtert Hospital, Milwaukee, Wisconsin
- Italy (2):
  - Ospedale Padiatrico Bambino Gesu Centro Fibrosi Cistica, Roma
  - Azienda Ospedaliera Universitaria Integrato di Verona Borgo Trento Centro Fibrosi Cistica, Verona
- United Kingdom (7):
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Ninewells Hospital Scottish Adult Cystic Fibrosis Service, Dundee
  - Western General Hospital Edinburgh, CF Adults / CF Unit, Edinburgh
  - NHS GGC, Glasgow
  - Raigmore Hospital, Inverness
  - St. James University Hospital, Leeds
  - Royal Victoria Infirmary Adult CF Centre, Newcastle upon Tyne

REFERENCES:
- [Derived] Devereux G, Wrolstad D, Bourke SJ, Daines CL, Doe S, Dougherty R, Franco R, Innes A, Kopp BT, Lascano J, Layish D, MacGregor G, Murray L, Peckham D, Lucidi V, Lovie E, Robertson J, Fraser-Pitt DJ, O'Neil DA. Oral cysteamine as an adjunct treatment in cystic fibrosis pulmonary exacerbations: An exploratory randomized clinical trial. PLoS One. 2020 Dec 28;15(12):e0242945. doi: 10.1371/journal.pone.0242945. eCollection 2020. PMID 33370348
- See also: NovaBiotics Website — http://www.novabiotics.co.uk/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 91 adult CF patients experiencing a pulmonary exacerbation were enrolled across 15 US and EU centres. 89 patients were randomised and 78 completed the 14 day treatment period of the study. First Patient first visit was 12 Jan 2017 and Last Patient last visit was 11 April 2018.
Pre-assignment Details: Of the 91 patients enrolled 89 patients met the inclusion criteria and 2 were not eligible:
  1 patient had <4 Fuchs criteria (not considered to be exacerbating)
  1 patient had reproductive issues
Groups:
- 450mg, Once Per Day: Patient takes one oral dose of Cysteamine (450mg) per day, in the morning. The patient takes two oral placebo doses, one at mid-day and one in the evening.
  Cysteamine: Oral Cysteamine Capsule
  Placebo Oral Capsule: Placebo Oral Capsule
- 150mg, Three Times Per Day: Patient takes three oral doses of Cysteamine (150mg) per day, one in the morning, one at mid-day and one in the evening.
  Cysteamine: Oral Cysteamine Capsule
  Placebo Oral Capsule: Placebo Oral Capsule
- 450mg, Twice Per Day: Patient takes two oral doses of Cysteamine (450mg) per day, one in the morning and one in the evening. The patient takes one oral placebo dose, at mid-day.
  Cysteamine: Oral Cysteamine Capsule
  Placebo Oral Capsule: Placebo Oral Capsule
- 300mg, Three Times Per Day: Patient takes three oral doses of Cysteamine (300mg) per day, one in the morning, one at mid-day and one in the evening.
  Cysteamine: Oral Cysteamine Capsule
  Placebo Oral Capsule: Placebo Oral Capsule
- 450mg, Three Times Per Day: Patient takes three oral doses of Cysteamine (450mg) per day, one in the morning, one at mid-day and one in the evening.
  Cysteamine: Oral Cysteamine Capsule
Period: Overall Study
Arm/Group | Placebo | 450mg, Once Per Day | 150mg, Three Times Per Day | 450mg, Twice Per Day | 300mg, Three Times Per Day | 450mg, Three Times Per Day
Started | 17 | 11 | 15 | 15 | 16 | 15
Day 14 Treatment Period | 17 | 10 | 13 | 14 | 13 | 14
Completed | 14 | 7 | 11 | 12 | 11 | 13
Not Completed | 3 | 4 | 4 | 3 | 5 | 2
Not completed — Adverse Event | 1 | 1 | 1 | 1 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Consent | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Failure to expectorate sputum | 1 | 0 | 1 | 0 | 1 | 0
Not completed — No gram negative | 1 | 2 | 1 | 1 | 1 | 1
Not completed — Patient had no transport | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Dosing | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- 450mg, Three Times Per Day: Patient takes three oral doses of Cysteamine (150mg) per day, one in the morning, one at mid-day and one in the evening.
  Cysteamine: Oral Cysteamine Capsule
- Total: Total of all reporting groups
Arm/Group | Placebo | 450mg, Once Per Day | 150mg, Three Times Per Day | 450mg, Twice Per Day | 300mg, Three Times Per Day | 450mg, Three Times Per Day | Total
Number analyzed (Participants) | 17 | 11 | 15 | 15 | 16 | 15 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.2 (5.64) | 27.5 (6.77) | 32.5 (12.7) | 32.3 (9.78) | 31.4 (12.0) | 27.5 (7.89) | 29.8 (9.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 5 | 8 | 8 | 8 | 43
  Male | 9 | 5 | 10 | 7 | 8 | 7 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 15 | 10 | 13 | 12 | 15 | 13 | 78
  Unknown or Not Reported | 2 | 1 | 2 | 2 | 1 | 2 | 10
BMI [Mean (Standard Deviation); unit: kg/m^2] | 20.2 (2.23) | 20.3 (3.03) | 20.7 (2.41) | 21.5 (2.21) | 20.5 (3.03) | 21.7 (2.84) | 20.8 (2.61)
Age at CF Diagnosis [Mean (Standard Deviation); unit: years] — Age at CF diagnosis was calculated as the date of CF diagnosis-date of birth
  years | 0.9 (2.41) | 3.9 (0.24) | 0.3 (0.49) | 1.6 (4.93) | 4.8 (11.45) | 1.8 (5.63) | 0.9 (2.41)
Duration of CF years [Mean (Standard Deviation); unit: years] — Duration of CF was calculated as the informed consent date - the date of diagnosis/365.25
  years | 26.36 (5.69) | 23.7 (9.26) | 32.45 (12.44) | 31.11 (10.92) | 26.76 (11.69) | 25.88 (7.07) | 27.85 (9.97)
FEV1 Percent predicted (%) [Mean (Standard Deviation); unit: litres per second] | 41.5 (15.31) | 39.4 (19.81) | 48.0 (18.26) | 46.1 (22.75) | 37.7 (13.44) | 46.9 (20.58) | 43.3 (18.34)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Sputum Bacterial Load
Description: Change from baseline through to Day 21 in log10 cfu/ml transformed total gram negative sputum bacterial load
Time Frame: Baseline through Day 21/End of Study
Population: Intention to treat population
Measure: Mean (Standard Deviation); unit: log 10 cfu/ml
Groups:
- 150mg, Three Times Per Day: Patient takes three oral doses of Cysteamine (l150mg) per day, one in the morning, one at mid-day and one in the evening.
  Cysteamine: Oral Cysteamine Capsule
  Placebo Oral Capsule: Placebo Oral Capsule
Arm/Group | Placebo | 450mg, Once Per Day | 150mg, Three Times Per Day | 450mg, Twice Per Day | 300mg, Three Times Per Day | High Dose, Three Times Per Day
Number analyzed (Participants) | 17 | 11 | 15 | 15 | 16 | 15
log 10 cfu/ml
  Day 7 change from baseline: number analyzed (Participants) | 17 | 9 | 13 | 12 | 10 | 14
  Day 7 change from baseline | -2.1 (2.887) | -1.03 (3.124) | -1.28 (1.978) | -1.7 (2.439) | -1.03 (1.997) | -0.25 (2.228)
  Day 14 change from baseline: number analyzed (Participants) | 15 | 10 | 12 | 11 | 10 | 15
  Day 14 change from baseline | -1.38 (2.291) | 0.12 (2.045) | -1.24 (2.686) | -1.32 (2.298) | -0.98 (1.894) | 0.33 (2.270)
  Day 21 change from baseline: number analyzed (Participants) | 14 | 10 | 13 | 12 | 10 | 13
  Day 21 change from baseline | -0.18 (1.238) | -1.22 (2.760) | -0.26 (1.639) | -1.04 (2.891) | -0.87 (1.677) | 0.93 (2.348)

2. Primary Outcome: Safety and Tolerability Assessed by the Number of Subjects With Adverse Events
Description: Assessed by variables such as adverse events (AEs), laboratory assessments, physical examinations, and vital signs.
Time Frame: Baseline through Day 21/End of Study
Population: Summary of participant reported adverse events (AEs) by study group
Measure: Number; unit: participants
Arm/Group | Placebo | 450mg, Once Per Day | 150mg, Three Times Per Day | 450mg, Twice Per Day | 300mg, Three Times Per Day | 450mg, Three Times Per Day
Number analyzed (Participants) | 17 | 11 | 15 | 15 | 16 | 15
participants
  Number of AEs | 30 | 29 | 40 | 33 | 45 | 36
  Number of SAEs | 1 | 1 | 2 | 1 | 0 | 1
  1 or more AEs | 9 | 10 | 11 | 12 | 10 | 13
  Severity of AE mild | 7 | 6 | 5 | 6 | 4 | 7
  Severity of AE moderate | 2 | 4 | 6 | 5 | 5 | 6
  Severity of AE severe | 0 | 0 | 0 | 1 | 1 | 0
  AEs leading to drug discontinuation | 1 | 1 | 1 | 1 | 1 | 1
  Nausea | 0 | 3 | 5 | 3 | 5 | 3
  Vomiting | 0 | 2 | 2 | 2 | 2 | 1
  Insomnia | 0 | 0 | 2 | 0 | 1 | 2
  Rash | 0 | 0 | 1 | 1 | 3 | 0
  Arthralgia | 0 | 1 | 1 | 1 | 0 | 1
  Decreased appetite | 0 | 0 | 1 | 0 | 2 | 1
  Haemoptysis | 2 | 0 | 1 | 1 | 2 | 0
  Oropharyngeal pain | 0 | 1 | 1 | 0 | 1 | 1
  Abdominal pain | 1 | 0 | 1 | 0 | 2 | 0
  Breath odour | 0 | 0 | 0 | 1 | 0 | 2

3. Secondary Outcome: Change From Baseline in Neutrophil Elastase Levels
Description: Actual values and change from baseline in neutrophil elastase levels were summarized using descriptive statistics by visit for each treatment group and each TDD group for the ITT Population.
Time Frame: Baseline through Day 21/End of Study
Population: Neutrophil Elastase Levels by Visit - Covariate Adjusted ANCOVA with Observed Data ITT Population
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- 450mg, Three Times Per Day: Patient takes three oral doses of Cysteamine 450mg) per day, one in the morning, one at mid-day and one in the evening.
  Cysteamine: Oral Cysteamine Capsule
Arm/Group | Placebo | 450mg, Once Per Day | 150mg, Three Times Per Day | 450mg, Twice Per Day | 300mg, Three Times Per Day | 450mg, Three Times Per Day
Number analyzed (Participants) | 17 | 11 | 15 | 15 | 16 | 15
ng/mL
  Day 7 change from baseline: number analyzed (Participants) | 15 | 10 | 12 | 14 | 12 | 14
  Day 7 change from baseline | -4659 (38335) | 23431 (53111) | 704 (36395) | -19623 (35548) | -15769 (40899) | 5135 (27791)
  Day 14 change from baseline: number analyzed (Participants) | 13 | 11 | 15 | 15 | 16 | 15
  Day 14 change from baseline | -3706 (42879) | -380 (157122) | -7208 (19210) | -12014 (23269) | -14083 (41215) | 14660 (35539)
  Day 21 change from baseline: number analyzed (Participants) | 13 | 10 | 13 | 11 | 12 | 14
  Day 21 change from baseline | -1000 (59856) | 4853 (18616) | 171 (19229) | -21002 (2472) | -14591 (39179) | -2558 (20068)

4. Secondary Outcome: Change From Baseline in Sputum IL8
Description: Sputum IL-8 Levels by Visit - Covariate Adjusted ANCOVA with Observed Data ITT Population
Time Frame: Baseline through Day 21/End of Study
Population: ITT Population
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | 450mg, Once Per Day | 150mg, Three Times Per Day | 450mg, Twice Per Day | 300mg, Three Times Per Day | 450mg, Three Times Per Day
Number analyzed (Participants) | 17 | 11 | 15 | 15 | 16 | 15
pg/mL
  Day 7 change from baseline | -26088 (55506) | -17864 (33785) | -5511 (46204) | 111574 (70338) | -2663 (41802) | -25785 (53721)
  Day 14 Change from baseline: number analyzed (Participants) | 13 | 10 | 10 | 11 | 12 | 13
  Day 14 Change from baseline | -28856 (39456) | -26528 (46737) | -33653 (55302) | 3167 (28204) | -6136 (53611) | 221 (30639)
  Day 21 change from baseline | 9576 (66157) | -16043 (34551) | -19778 (49306) | 2831 (23050) | 631 (32350) | -10671 (65656)

5. Secondary Outcome: Change From Baseline in FEV1
Description: Change from Baseline in FEV1 Percent Predicted (%) - Covariate Adjusted ANCOVA with Observed Data ITT Population
Time Frame: Baseline through Day 21/End of Study
Population: Change from Baseline in FEV1 Percent Predicted (%) - Covariate Adjusted ANCOVA with Observed Data ITT Population
Measure: Mean (Standard Deviation); unit: percentage of predicted
Arm/Group | Placebo | 450mg, Once Per Day | 150mg, Three Times Per Day | 450mg, Twice Per Day | 300mg, Three Times Per Day | 450mg, Three Times Per Day
Number analyzed (Participants) | 17 | 11 | 15 | 15 | 16 | 15
percentage of predicted
  Day 7 change from baseline: number analyzed (Participants) | 17 | 10 | 13 | 15 | 14 | 15
  Day 7 change from baseline | 7.9 (13.67) | 4.4 (5.52) | 6.9 (8.85) | 11.8 (9.96) | 4.9 (5.48) | 3.7 (8.65)
  Day 14 change from baseline: number analyzed (Participants) | 17 | 10 | 13 | 14 | 13 | 14
  Day 14 change from baseline | 9.2 (14.03) | 4.0 (5.14) | 8.9 (10.87) | 13.6 (10.83) | 5.3 (6.65) | 7.5 (7.07)
  Day 21 change from baseline: number analyzed (Participants) | 16 | 10 | 13 | 14 | 13 | 14
  Day 21 change from baseline | 9.5 (13.5) | 4.7 (5.03) | 6.5 (7.25) | 8.9 (10.66) | 6.4 (8.18) | 6.3 (11.34)

6. Secondary Outcome: Change From Baseline in BMI
Description: BMI (kg/m^2) by Visit - ANCOVA with Observed Data ITT Population
Time Frame: Baseline through Day 21/End of Study
Population: ITT
Measure: Mean (Standard Deviation); unit: kg/m^2 for BMI
Arm/Group | Placebo | 450mg, Once Per Day | 150mg, Three Times Per Day | 450mg, Twice Per Day | 300mg, Three Times Per Day | 450mg, Three Times Per Day
Number analyzed (Participants) | 17 | 11 | 15 | 15 | 16 | 15
kg/m^2 for BMI
  BMI Day 7 change from baseline: number analyzed (Participants) | 16 | 10 | 13 | 15 | 13 | 15
  BMI Day 7 change from baseline | 0.39 (0.371) | 0.32 (0.498) | 0.28 (0.3) | 0.24 (0.428) | 0.15 (0.586) | 0.15 (0.589)
  BMI Day 14 change from baseline: number analyzed (Participants) | 16 | 10 | 13 | 14 | 12 | 14
  BMI Day 14 change from baseline | 0.34 (0.452) | 0.64 (0.505) | 0.34 (0.477) | 0.37 (0.488) | 0.23 (0.705) | 0.32 (0.893)
  BMI Day 21 change from baseline: number analyzed (Participants) | 15 | 10 | 13 | 14 | 11 | 14
  BMI Day 21 change from baseline | 0.54 (0.537) | 0.55 (0.553) | 0.47 (0.564) | 0.18 (0.478) | -0.02 (0.980) | 0.12 (0.828)

7. Secondary Outcome: Change From Baseline in C-Reactive Protein
Description: Change from baseline in C-Reactive Protein at visits 7, 14 and 21
Time Frame: Baseline through Day 21
Population: CRP by visit ANCOVA with observed data ITT population
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Placebo | 450mg, Once Per Day | 150mg, Three Times Per Day | 450mg, Twice Per Day | 300mg, Three Times Per Day | 450mg, Three Times Per Day
Number analyzed (Participants) | 17 | 11 | 15 | 15 | 16 | 15
nmol/L
  Day 7 change from baseline: number analyzed (Participants) | 17 | 10 | 13 | 15 | 12 | 15
  Day 7 change from baseline | -182.828 (188.1222) | -285.006 (295.0114) | -229.821 (590.1267) | -318.933 (344.9138) | -120.193 (200.2307) | -281.752 (293.2595)
  Day 14 change from baseline: number analyzed (Participants) | 15 | 10 | 13 | 14 | 12 | 14
  Day 14 change from baseline | -75.671 (331.2220) | -312.435 (323.8782) | -216.105 (617.1174) | -215.242 (225.7293) | -111.272 (124.8394) | -294.13 (509.9255)
  Day 21 change from baseline: number analyzed (Participants) | 14 | 10 | 13 | 14 | 12 | 14
  Day 21 change from baseline | -44.341 (296.4493) | -237.062 (378.4493) | -116.442 (730.9709) | -198.759 (235.0256) | -23.421 (157.4203) | -225.787 (543.1070)

8. Secondary Outcome: Change From Baseline in Blood Leukocyte Count
Description: Blood Leukocyte Count (10^9 leucocytes/L) by Visit - ANCOVA with Observed Data ITT Population
Time Frame: Baseline through Day 21/End of Study
Population: ITT
Measure: Mean (Standard Deviation); unit: 10^9 leucocytes/L
Arm/Group | Placebo | 450mg, Once Per Day | 150mg, Three Times Per Day | 450mg, Twice Per Day | 300mg, Three Times Per Day | 450mg, Three Times Per Day
Number analyzed (Participants) | 17 | 11 | 15 | 15 | 16 | 15
10^9 leucocytes/L
  Day 7 change from baseline: number analyzed (Participants) | 16 | 10 | 13 | 13 | 13 | 15
  Day 7 change from baseline | -2.553 (4.617) | -1.836 (2.0566) | -2.808 (3.595) | -2.482 (3.4502) | -2.575 (3.1189) | -2.863 (2.9932)
  Day 14 change from baseline: number analyzed (Participants) | 15 | 10 | 12 | 14 | 12 | 14
  Day 14 change from baseline | -1.568 (4.7176) | -2.220 (2.3451) | -2.648 (3.9122) | -3.419 (3.5734) | -0.193 (3.8376) | -4.066 (2.4102)
  Day 21 change from baseline: number analyzed (Participants) | 14 | 10 | 13 | 14 | 12 | 14
  Day 21 change from baseline | -1.870 (4.6187) | -1.757 (2.6670) | -1.880 (3.0935) | -1.763 (3.3193) | -0.127 (2.5869) | -3.316 (3.6322)

9. Secondary Outcome: Assessment of Blood Cysteamine Levels
Description: Study Drug Plasma at Day 14 Safety Population
Time Frame: Day 14
Population: Safety population
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Placebo | 450mg, Once Per Day | 150mg, Three Times Per Day | 450mg, Twice Per Day | 300mg, Three Times Per Day | 450mg, Three Times Per Day
Number analyzed (Participants) | 15 | 10 | 13 | 14 | 12 | 14
ng/ml | 10.0 (0.00) | 515.11 (683.956) | 102.45 (144.863) | 347.76 (507.747) | 256.85 (377.262) | 256.84 (251.593)

10. Secondary Outcome: Assessment of Sputum Cysteamine Levels
Description: Study Drug Sputum Concentrations at Day 14 Safety Population
Time Frame: Day 14
Population: Safety Population - there are fewer numbers of patients due to the inability of some patients to provide sputum samples
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Placebo | 450mg, Once Per Day | 150mg, Three Times Per Day | 450mg, Twice Per Day | 300mg, Three Times Per Day | 450mg, Three Times Per Day
Number analyzed (Participants) | 15 | 9 | 10 | 10 | 12 | 14
ng/ml | 150.0 (0.00) | 682.8 (1009.8) | 150.0 (0.0) | 316.4 (1423.6) | 739.7 (1423.6) | 811.1 (917.49)

11. Secondary Outcome: Change From Baseline in CFRSD-CRISS
Description: Mean Change from Baseline in Cystic Fibrosis Respiratory Symptom Diary (CFRSD)-Chronic Respiratory Infection Symptom Scale (CRISS) CRFSD-CRISS:The CFRSD is a 16-item PROM to evaluate the effect of treatment on the severity of symptoms of acute respiratory infections associated with CF (i.e., CFRSD-CRISS) and to assess the emotional and activity impacts of these symptoms. The overall CRISS score range is 0-100 with 100 being the most severe symptoms.The CFRSD-CRISS is a validated unidimensional scale based on a subset of 8 items from the CFRSD questionnaire that quantifies symptom severity for the previous 24 hours to capture the magnitude of symptoms in stable CF, during medically treated CF exacerbations, and during recover from an exacerbation. The 8 items on the CFRSD-CRISS were scored using a 5-point Likert scale ranging from 0 (no symptom) to 4 (the highest magnitude of severity). So score range of 0-32.
Time Frame: Baseline through to Day 21
Population: Mean Change from Baseline in CRFSD-CRISS - Linear MMRM Model with Observed Data (ITT Population)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 450mg, Once Per Day | 150mg, Three Times Per Day | 450mg, Twice Per Day | 300mg, Three Times Per Day | 450mg, Three Times Per Day
Number analyzed (Participants) | 17 | 11 | 15 | 15 | 16 | 15
units on a scale
  Day 7 change from baseline: number analyzed (Participants) | 17 | 10 | 13 | 15 | 14 | 15
  Day 7 change from baseline | -16.4 (8.31) | -18.1 (10.19) | -11.9 (7.98) | -19.1 (10.65) | -10.5 (5.91) | -17.8 (12.67)
  Day 14 change from baseline: number analyzed (Participants) | 17 | 10 | 13 | 14 | 13 | 14
  Day 14 change from baseline | -16.3 (15.0) | -24.3 (16.35) | -15.5 (12.48) | -28.1 (16.88) | -14.8 (8.53) | -23.9 (16.41)
  Day 21 change from baseline | -18.3 (11.7) | -23.2 (13.36) | -15.8 (11.68) | -19.9 (19.23) | -12.9 (6.37) | 22.0 (17.71)

12. Secondary Outcome: Change From Baseline in CFQ-R
Description: The CFQ-R is a disease-specific HRQOL (Health related quality of life) measure containing both generic and CF-specific scales and measures functioning during the previous 2 weeks. Each CFQ-R scale yielded standardized scores ranging from 0 to 100; higher scores indicated better HRQOL
Time Frame: Baseline through Day 21/End of Study
Population: Change from Baseline to Day 14 in CFQ-R Respiratory Score: ANCOVA with Observed Data ITT Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 450mg, Once Per Day | 150mg, Three Times Per Day | 450mg, Twice Per Day | 300mg, Three Times Per Day | 450mg, Three Times Per Day
Number analyzed (Participants) | 17 | 11 | 15 | 15 | 16 | 15
units on a scale
  Day 7 Change from baseline: number analyzed (Participants) | 17 | 10 | 13 | 15 | 14 | 15
  Day 7 Change from baseline | 14.7 (18.21) | 12.2 (13.81) | 12.0 (16.32) | 12.1 (14.95) | 15.9 (14.1) | 19.6 (16.11)
  Day 14 change from baseline: number analyzed (Participants) | 17 | 10 | 13 | 14 | 13 | 14
  Day 14 change from baseline | 22.9 (21.51) | 24.4 (14.15) | 19.7 (16.76) | 31.3 (17.38) | 21.8 (14.07) | 28.6 (15.69)
  Day 21 change from baseline: number analyzed (Participants) | 16 | 10 | 13 | 14 | 13 | 14
  Day 21 change from baseline | 24.3 (19.34) | 30.6 (17.62) | 25.2 (19.19) | 31.3 (30.08) | 24.8 (14.85) | 37.3 (23.61)

13. Secondary Outcome: Change From Baseline in Jarad and Sequeiros Symptom Score Questionnaire
Description: The Jarad and Sequeiros Symptom Questionnaire (Jarad, 2012) is a simple participant-completed questionnaire that assesses and evaluates change in participant symptoms related to different aspects of respiratory function during a CF exacerbation. The questionnaire consists of 4 questions, each answered on a 4-point scale ranging from 1 (best) to 4 (worst). A range of minimum 4 to maximum16.Jarad and Sequeiros Questionnaire Score - changes from baseline at day 7 and day 14
Time Frame: changes from baseline at day 7 and day 14
Population: ITT Linear MMRM Model with Observed Data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 450mg, Once Per Day | 150mg, Three Times Per Day | 450mg, Twice Per Day | 300mg, Three Times Per Day | 450mg, Three Times Per Day
Number analyzed (Participants) | 17 | 11 | 15 | 15 | 16 | 15
units on a scale
  change from baseline to day 7: number analyzed (Participants) | 17 | 10 | 13 | 15 | 14 | 15
  change from baseline to day 7 | -2.6 (1.97) | -1.9 (2.38) | -1.4 (1.85) | -3.3 (2.35) | -2.4 (2.21) | -3.1 (3.33)
  change from baseline to day 14: number analyzed (Participants) | 17 | 10 | 13 | 14 | 13 | 14
  change from baseline to day 14 | -3.2 (2.9) | -2.9 (2.6) | -2.0 (2.48) | -4.3 (2.16) | -3.1 (2.63) | -4.2 (3.19)

14. Secondary Outcome: Change From Baseline in Weight
Description: Weight (kg) by visit - ANCOVA with observed data
Time Frame: Baseline through Day 21/End of Study
Population: ITT
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Placebo | 450mg, Once Per Day | 150mg, Three Times Per Day | 450mg, Twice Per Day | 300mg, Three Times Per Day | 450mg, Three Times Per Day
Number analyzed (Participants) | 17 | 11 | 15 | 15 | 16 | 15
kg
  Day 7: number analyzed (Participants) | 17 | 10 | 13 | 15 | 14 | 15
  Day 7 | 0.96 (1.084) | 0.83 (1.241) | 0.79 (1.145) | 0.67 (1.182) | 0.25 (1.547) | 0.36 (1.74)
  Day 14: number analyzed (Participants) | 17 | 10 | 13 | 14 | 13 | 14
  Day 14 | 0.85 (1.355) | 1.71 (1.270) | 0.96 (1.368) | 1.04 (1.445) | 0.55 (1.872) | 0.89 (2.621)
  Day 21: number analyzed (Participants) | 16 | 10 | 13 | 14 | 12 | 14
  Day 21 | 1.37 (1.486) | 1.50 (1.639) | 1.30 (1.503) | 0.52 (1.295) | -0.28 (2.728) | 0.34 (2.477)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline (day 0, day study treatment commences) until day 21 (end of study/follow up)
Description: An AE was defined as any untoward medical occurrence in a participant in a clinical investigation who was administered a pharmaceutical product. The AE did not necessarily have a causal relationship with this product. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the investigational product, whether or not related to the investigational product.
Arm/Group | Placebo | High Dose, Once Per Day | Low Dose, Three Times Per Day | High Dose, Twice Per Day | Mid-Range Dose, Three Times Per Day | High Dose, Three Times Per Day
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/11 | 0/15 | 0/15 | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/17 | 1/11 | 2/15 | 1/15 | 0/16 | 1/15
Other Adverse Events (participants affected / at risk) | 9/17 | 10/11 | 11/15 | 12/15 | 10/16 | 13/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=17) | High Dose, Once Per Day (N=11) | Low Dose, Three Times Per Day (N=15) | High Dose, Twice Per Day (N=15) | Mid-Range Dose, Three Times Per Day (N=16) | High Dose, Three Times Per Day (N=15)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Prolongation of hospitalisation
Axillary vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Right axillary deep vein thrombosis
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Kidney Stone
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Depression exacerbation manifesting in suicidal and homicdal ideation
Infective pulmonary exacerbation of CF (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Pulmonary exacerbation hospitalisation prolongation of hospitalisation
Campylobacter sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Campylobacter septicaemia hospitalisation prolongation of hospitalisation
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=17) | High Dose, Once Per Day (N=11) | Low Dose, Three Times Per Day (N=15) | High Dose, Twice Per Day (N=15) | Mid-Range Dose, Three Times Per Day (N=16) | High Dose, Three Times Per Day (N=15)
Nausea (Gastrointestinal disorders) | 0/0 (0) | 3 (3) | 5 (5) | 3 (3) | 5 (5) | 3 (3)
vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breath odour (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingival recession (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-tussive vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 5 (5) | 1 (1) | 3 (3) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysguesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Intention tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sinus Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
pyrexia (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Administration site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adminstration site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Crepitations (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sensation of foreign body (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection (bacterial) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Campylobacter sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficle colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficle infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth abcess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary function test decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carbon dioxide (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonoscopy (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eosinophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mycobacterium tuberculosis complex test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Dermatitis allergic (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Axillary vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion site reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stoma site reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oligomenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-18): https://cdn.clinicaltrials.gov/large-docs/48/NCT03000348/Prot_SAP_000.pdf